CLINICAL TRIAL: NCT06610682
Title: Feasibility of CSF (Cerebrospinal Fluid) and Plasma ctDNA (Circulating Tumor Deoxyribonucleic) in BRAF (V-raf Murine Sarcoma Viral Oncogene Homolog B1)-Altered Glioma During Treatment With Plixorafenib
Brief Title: Feasibility of CSF and Plasma ctDNA in BRAF-altered Glioma During Treatment With Plixorafenib
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Fore Biotherapeutics (Industry); Ivy Brain Tumor Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2488; Foundatin (Other: Ivy Foundation); IRB00457005 (Other: Johns Hopkins Medicine IRB)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: BRAF V600E Mutation
Keywords: BRAF,; BRAF V600E mutant; Plixorafenib
MeSH Terms: interventions — Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Recurrent BRAF-V600E mutant gliomas previously received BRAFi* +/- MEKi** , (Experimental): *BRAFi (v-raf murine sarcoma viral oncogene homolog B1 inhibitor)
  **MEKi (Methyl ethyl ketone inhibitor)
  Interventions: Drug: Plixorafenib; Drug: Cobicistat 150 MG [Tybost]

INTERVENTIONS:
Drug: Plixorafenib — Plixorafenib (900mg) daily co-administered with cobicistat (150mg daily) 7-28 days post-operatively, when clinically stable. Patients will take the drug daily by mouth under fasting conditions continuously for 28-day cycles until progressive disease or up to 24 cycles
Drug: Cobicistat 150 MG [Tybost] — Plixorafenib (900mg) daily co-administered with cobicistat (150mg daily) 7-28 days post-operatively, when clinically stable. Patients will take the drug daily by mouth under fasting conditions continuously for 28-day cycles until progressive disease or up to 24 cycles

SUMMARY:
Evaluating the sensitivity and feasibility of using ctDNA assays optimized for detecting very low ctDNA counts from cerebrospinal fluid (CSF) and plasma. The investigators will evaluate the sensitivity of ctDNA from plasma and CSF at baseline (defined as Cycle1 Day1 (C1D1) pre-treatment) and over time in response to treatment with plixorafenib co-administered with cobicistat in BRAF-V600E mutant glioma refractory to prior therapies.

DETAILED DESCRIPTION:
This clinical trial is designed as a pilot, signal-finding study to demonstrate the feasibility of detecting ctDNA at baseline and after 4 weeks of treatment (primary endpoint), as well as correlating with disease status as per radiographic response (RR; secondary endpoint). In addition, the investigators will generate preliminary data for activity of plixorafenib co-administered with cobicistat in this heavily-pretreated population. Patients with measurable (by Response Assessment in Neuro-Oncology (RANO 2.0)), recurrent BRAF-V600E mutant glioma will be screened and consented for the study prior to surgery. Patients will undergo pre-operative MRI and clinically-indicated resection or biopsy (specific approach as per treating neurosurgeon) for confirmation of progression and characterization of potential acquired resistance alterations. All patients will have a ventricular reservoir placed at time of surgery with CSF and plasma sampling. Patients will start the study drug (plixorafenib 900mg daily co-administered with cobicistat 150mg daily) 7-28 days post-operatively, when clinically stable. Patients will take the drug daily by mouth under fasting conditions continuously for 28-day cycles until progressive disease or up to 24 cycles. MRI will be performed post-operatively (between proof of delivery (POD#0) and start of study drug) for evaluation of measurable disease, after Cycle 1, then every 2 cycles. Blood and CSF samples will be obtained on day of surgery, at baseline, pre-C2, then with each MRI. A total of 12 evaluable patients will be enrolled. Patients who do not start drug will be replaced, up to a total of 15 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of a primary central nervous system (CNS) tumor with documented BRAF-V600E mutation by a Clinical Laboratory Improvement Amendments (CLIA) approved DNA or RNA (Ribonucleic acid )-based sequencing test (NGS (Next generation sequencing) or RNAseq). Immunohistochemistry alone is insufficient.
2. Patient must have received prior BRAF and/or Mitogen-activated protein kinase kinase (MEK) inhibitor therapy.
3. Karnofsky performance status ≥ 70.
4. Patient is 18 years of older.
5. Measurable disease by RANO2.0 criteria on screening MRI. Leptomeningeal disease allowed.
6. Willing to submit archival tumor sample if available.
7. The following intervals from previous treatments should have elapsed prior to cycle 1 day 1:

   * 12 weeks from the completion of radiation.
   * 12 weeks from an anti- vascular endothelial growth factor therapy (VEGF)
   * 4 weeks from a nitrosourea chemotherapy
   * 3 weeks from a non-nitrosourea chemotherapy
   * 2 weeks or 5 half-lives from any investigational (not FDA-approved) agents (whichever is shorter)
   * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., erlotinib, hydroxychloroquine, dabrafenib, etc.)
8. Patients must have the following organ and marrow function:

   * Absolute neutrophil count >1,000/micro liter (mcL)
   * Platelets >100,000/mcL
   * Hemoglobin > 9 g/dL
   * Total bilirubin </= 1.5 x institutional upper limit of normal (ULN) OR total bilirubin >1.5 × ULN with direct bilirubin <1.5 × ULN
   * (aspartate aminotransferase (AST) and alanine transaminase (ALT) </= 2.5 x institutional ULN
   * prothrombin time (PT) or Partial thromboplastin time (PTT) < 1.5 x institutional ULN
   * Creatinine ≤ 1.5 x institutional ULN OR Creatinine clearance (Cockcroft-Gault Formula) > 50 ml/min/1.73m2
9. Patient must be able to provide written informed consent.
10. All adverse events related to prior therapies (chemotherapy; radiotherapy; surgery) must have resolved to Grade 1 or baseline except for

    * Alopecia (Grade ≤2)
    * Sensory neuropathy (Grade ≤2)
    * Lymphopenia (Grade 2)
    * Other adverse events that have resolved to Grade ≤2 that, according to the clinical judgment of the investigator, do not constitute a safety risk to the participant.
11. Patients must be maintained on a stable or decreasing dose of systemic corticosteroid regimen (no increase for 5 days) prior to screening MRI. Topical and inhaled steroid treatment is allowed.
12. Ability to swallow and retain orally administered medications, including a liquid suspension.
13. Female participants of childbearing potential must have a negative serum pregnancy test prior to study start. Female participants of childbearing potential must agree to use highly effective contraception and not to donate ova from screening through 30 days after the last dose of study drug. Highly effective contraception is defined as 1) intrauterine device, 2) abstinence, or 3) combined estrogen and progesterone or progesterone only containing implants, injectables, transdermal, or intravaginal contraceptives. Male participants must also agree to use adequate contraception and not to donate sperm from screening until 90 days after the last dose of study drug.
14. Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder. Patients with other malignancies must be disease-free for >/=2 years.
15. Life expectancy equal or greater than six months.

Exclusion Criteria:

1. Current use of any other standard or investigational agents (excepting tumor treating fields).
2. Known co-occurring NF-1 (Neurofibromatosis type 1) and/or reticular activating system (RAS) -related alteration known to cause resistance.
3. Prior treatment with any rapidly accelerated fibrosarcoma (RAF) dimer disruptor or pan-RAF inhibitor.
4. Known hypersensitivity to plixorafenib, cobicistat or excipients.
5. Current use of a prohibited medication (including herbal medications, supplements, or foods), as described in Section 5.6, or use of a prohibited medication ≤ 7 days prior to surgery date.
6. Impairment in gastrointestinal function or disease that may significantly alter the absorption of oral plixorafenib or cobicistat (such as ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
7. Clinically significant cardiovascular disease including, but not limited to the following:

   * History of acute coronary syndromes (including myocardial infarction or unstable angina), coronary artery bypass grafting, coronary angioplasty or stenting ≤ 180 days prior to start date;
   * Congestive heart failure requiring treatment (New York Heart Association Grade > 2);
   * History or presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia);
   * Corrected QT interval (QTcF) QT corrected for heart rate by Fridericia's cube root formula) interval ≥ 480 ms.
8. History of recent (≤ 90 days) thromboembolic or cerebrovascular event such as transient ischemic attack, cerebrovascular accident, or hemodynamically significant (massive or sub-massive) deep vein thrombosis or pulmonary emboli (DVT/PE). Note: Patients with DVT/PE that does not result in hemodynamic instability may enroll as long as participants are anticoagulated for at least 4 weeks. Note: Patients with Deep vein thrombosis (DVT)/pulmonary embolism (PE) related to indwelling catheters or other procedures may enroll.
9. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible.
10. Pregnant women are excluded from this study because the effects of plixorafenib on a fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with plixorafenib or cobicistat, breastfeeding should be discontinued if the mother is treated on study.
11. No contraindication to clinically-indicated surgery.
12. No contraindication to ventricular reservoir placement or biospecimen collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with ctDNA in CSF or plasma | 4 weeks
  Estimate detection rates of BRAF-V600 ctDNA from CSF and blood at A) baseline (defined as C1D1 pre-treatment) and B) week 4 after treatment.

SECONDARY OUTCOMES:
Compare BRAF-V600 ctDNA levels in CSF and plasma after treatment among patients with different radiographic responses | 12 weeks
  Compare BRAF-V600 ctDNA levels at baseline and week 4 after treatment among patients with different radiographic responses (1="improved", 2="stable", 3="worsened" measured by RANO2.0 criteria) at 4 and 12 weeks after the treatment initiation.

OTHER OUTCOMES:
Identify co-occurring genetic, epigenetic, or expression signatures correlating with response. | 12 weeks
  Co-occurring genetic, epigenetic, or expression signatures correlating with response.
Correlation of ctDNA levels with response | 2 years
  using Rano2.0 Criteria
Correlation of ctDNA levels with progression-free survival | 2 years
  Progression-free survival measured by the time from first treatment to disease progression or death
Correlation of ctDNA levels with overall survival. | 2 years
  time of first dose to death

CONTACTS AND LOCATIONS:
Overall Officials: Karisa Schreck, MD, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States